CLINICAL TRIAL: NCT04352790
Title: Multifactorial Risk Stratification in Patients With Ischemic Stroke or Transient Ischemic Attack and Structural, Inflammatory, or Arrhythmogenic Cardiac Disease
Brief Title: Multifactorial Risk Stratification in Stroke Patients With Cardiac Disease
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Other Study IDs: 402/2009BO2, 522/2012BO2
Record Dates: First submitted 2020-04-15; First posted 2020-04-20 (Actual); Last update posted 2020-04-22 (Actual); Status verified 2020-04

CONDITIONS: Stroke; Cardiac Disease
Keywords: patent foramen ovale; loop recorder; atrial fibrillation; heart rhythm monitoring; autonomic dysfunction; cryptogenic stroke; embolic stroke of undetermined source; ESUS; transient ischemic attack; retinal ischemia
MeSH Terms: conditions — Stroke; Heart Diseases; Foramen Ovale, Patent; Atrial Fibrillation; Primary Dysautonomias; Ischemic Stroke; Ischemic Attack, Transient

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Prospective registry for multifactorial risk factor assessment, enrolling consecutive ischemic stroke/transient ischemic attack patients with structural, inflammatory, or arrhythmogenic cardiac disease, who are admitted to our University Hospital.

DETAILED DESCRIPTION:
The prospective registry shall provide new insights into the multiple associations, and respective therapeutic implications of cardio-vascular risk factors and stroke. For that reason consecutive patients with ischemic stroke/transient ischemic attack (brain, spinal cord, or retinal) and structural (e.g. patent foramen ovale), septic or aseptic endocarditis or myocarditis, or supra-ventricular or ventricular arrhythmia, who are admitted to our University Hospital, are enrolled. Multifactorial assessment of risk factors is based on medical history, laboratory biomarkers, electrocardiogram incl. cardiac autonomic function analysis, and (long-term) cardiac rhythm monitoring, as well as transthoracic and transesophageal echocardiography. Inclusion of follow-up visits permit longitudinal and prognostic evaluation of routine diagnostic and therapeutic interventions for secondary stroke prevention (e.g. implantable loop recorders or interventional closure of patent foramen ovale).

ELIGIBILITY:
Inclusion Criteria:

* Ischemic stroke or transient ischemic attack (brain, spinal cord, or retinal)

Exclusion Criteria:

* Acute intracranial hemorrhage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive ischemic stroke/transient ischemic attack patients (brain, spinal crd, or retinal) with structural, inflammatory, or arrhythmogenic cardiac disease, who are admitted to our University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 878 (Actual)
Dates: Start 2012-03-01 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of any stroke | ≥ 12 months
  Recurrent ischemic stroke or intracranial hemorrhage during follow-up

SECONDARY OUTCOMES:
Rate of mortality | ≥ 12 months
  Death from any cause during follow-up
Rate of ischemic stroke | ≥ 12 months
  Ischemic stroke recurrence during follow-up
Rate of transient ischemic attack | ≥ 12 months
  Transient ischemic attack recurrence during follow-up
Rate of systemic embolism | ≥ 12 months
  Systemic embolism during follow-up
Rate of myocardial infarction | ≥ 12 months
  Myocardial infarction during follow-up
Rate of intracranial hemorrhage | ≥ 12 months
  Intracranial hemorrhage during follow-up
Rate of major Bleedings | ≥ 12 months
  Major Bleedings during follow-up
Rate of major or clinically relevant non-major bleedings | ≥ 12 months
  Major or clinically relevant non-major bleedings during follow-up
Rate of serious adverse events | ≥ 12 months
  Serious adverse events during follow-up
Rate of new-onset atrial fibrillation | ≥ 12 months
  Detection of atrial fibrillation during follow-up
modified Rankin Score; range from 0 to 6, with '0' indicating the best outcome (i.e. no deficit), and '6' the worst outcome (i.e. death) | ≥ 12 months
  modified Rankin Scale score at follow-up

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Poli S, Diedler J, Hartig F, Gotz N, Bauer A, Sachse T, Muller K, Muller I, Stimpfle F, Duckheim M, Steeg M, Eick C, Schreieck J, Gawaz M, Ziemann U, Zuern CS. Insertable cardiac monitors after cryptogenic stroke--a risk factor based approach to enhance the detection rate for paroxysmal atrial fibrillation. Eur J Neurol. 2016 Feb;23(2):375-81. doi: 10.1111/ene.12843. Epub 2015 Oct 16. PMID 26470854
- [Derived] Poli S, Siebert E, Mbroh J, Poli K, Krumbholz M, Mengel A, Greulich S, Hartig F, Muller KAL, Bocksch W, Gawaz M, Ziemann U, Zuern CS. Closure or medical therapy of patent foramen ovale in cryptogenic stroke: prospective case series. Neurol Res Pract. 2021 Apr 1;3(1):16. doi: 10.1186/s42466-021-00114-3. PMID 33789756